CLINICAL TRIAL: NCT00033358
Title: Modulation Of Putative Surrogate Endpoint Biomarkers In Endometrial Biopsies From Women With HNPCC
Brief Title: Hormone Therapy in Preventing Endometrial Cancer in Patients With a Genetic Risk For Hereditary Nonpolyposis Colon Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2013-00466; ID01-340; CDR0000069277; NCI-P02-0218; MDA-ID-01340; N01CN05127 (Other Grant/Funding Number: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Medroxyprogesterone; Medroxyprogesterone Acetate; Ethinyl Estradiol; Norgestrel; Levonorgestrel

ARMS (2):
- Arm I (medroxyprogesterone) (Experimental): Patients receive medroxyprogesterone intramuscularly once on day 1. Approximately 90 days after the injection, patients undergo a repeat transvaginal ultrasound and endometrial biopsy.
  Interventions: Drug: medroxyprogesterone; Other: laboratory biomarker analysis
- Arm II (ethinyl estradiol, norgestrel) (Experimental): Patients receive OCP comprising ethinyl estradiol and norgestrel once daily on days 1-21. Treatment repeats every 28 days for 3-4 courses (3-4 packs of OCP) in the absence of unacceptable toxicity. Approximately 1 week after starting the fourth pack of OCP, patients undergo a repeat transvaginal ultrasound and endometrial biopsy.
  Interventions: Drug: ethinyl estradiol; Drug: norgestrel; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: medroxyprogesterone — Given intramuscularly
  Other Names: Depo-Provera; medroxyprogesterone acetate; MPA; Provera; Provera Dosepak
  Arms: Arm I (medroxyprogesterone)
Drug: ethinyl estradiol — Given orally
  Other Names: Diogyn E; EE; Estinyl; Ethinoral; Eticylol
  Arms: Arm II (ethinyl estradiol, norgestrel)
Drug: norgestrel — Given orally
  Other Names: Microlut; NORGES; Ovrette; Wy-3707
  Arms: Arm II (ethinyl estradiol, norgestrel)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Randomized phase II trial to compare two different hormone therapy regimens in preventing endometrial cancer in women who have a genetic risk for hereditary nonpolyposis colon cancer. Hormone therapy may prevent the development of endometrial cancer in women with a genetic risk for hereditary nonpolyposis colon cancer. It is not yet known which hormone therapy regimen is more effective in preventing endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective is to evaluate the effect of progesterone therapy versus combination estrogen and progesterone therapy on potential surrogate endpoint biomarkers (SEBs) relevant to endometrial carcinogenesis.

II. To evaluate changes in histology and ultrasound appearance of the endometrium in women with HNPCC after 3 months of progesterone therapy versus combination estrogen and progesterone therapy compared with baseline.

III. To establish a point estimate of the baseline frequency of endometrial abnormalities looking at histological and molecular markers in a cohort of females carrying an HNPCC gene mutation.

OUTLINE: Patients are randomized to 1 of 2 arms.

All patients undergo a baseline transvaginal ultrasound and endometrial biopsy.

Arm I: Patients receive medroxyprogesterone intramuscularly once on day 1. Approximately 90 days after the injection, patients undergo a repeat transvaginal ultrasound and endometrial biopsy.

Arm II: Patients receive oral contraceptive pills (OCP) comprising ethinyl estradiol and norgestrel once daily on days 1-21. Treatment repeats every 28 days for 3-4 courses (3-4 packs of OCP) in the absence of unacceptable toxicity. Approximately 1 week after starting the fourth pack of OCP, patients undergo a repeat transvaginal ultrasound and endometrial biopsy.

Patients are followed at 6 weeks and are encouraged to return in 6 months to participate in continued endometrial screening.

ELIGIBILITY:
Inclusion Criteria:

* Women with known mutation of an HNPCC-associated gene (hMLH-1, hMSH-2, or hMSH-6) or fulfill Amsterdam Criteria and have had one or more HNPCC-associated cancers
* No prior hysterectomy; (participants may be scheduled for prophylactic hysterectomy following the study)
* Voluntary consent documented by a signed and witnessed informed consent
* Negative serum pregnancy test at baseline evaluation
* No history of pelvic irradiation for whatever cause
* No chemotherapy for two years
* Women >= 40 must have had a screening mammogram within the last 12 months prior to participation in this study
* Women who are at 50% risk of having a mutation and willing to have genetic testing

Exclusion Criteria:

* Use of oral contraceptives or depoMPA or hormonal exposure, such as hormonal IUD, tamoxifen, raloxifene, or other selective estrogen receptor modulators (SERMs) within four months of initiating study; women will be asked to be off oral contraceptives or other hormonal exposure for 4 months prior to initiating study
* Medical contraindication to use of oral contraceptives or depoMPA including:

  * Known or suspected pregnancy
  * Undiagnosed vaginal bleeding
  * Known or suspected malignancy of breast or endometrium
  * Active thrombophlebitis, or current or past history of thromboembolic disorders, or cerebral vascular disease
  * Gall bladder disease or liver dysfunction or disease, including hepatic adenomas or carcinoma, or abnormal liver function tests
  * Known hypersensitivity to depoMPA contraceptive injection (medroxyprogesterone acetate or any of its other ingredients)
  * Depression that is currently not under control, in the judgement of the Principal Investigator
  * History of epilepsy
  * History of diabetes
  * Coronary artery disease
  * Age >=35 and a current tobacco smoker
* Known inability to participate in the scheduled follow-up tests (i.e., alcohol dependence or illicit drug use)
* Significant medical history or psychiatric problems which would make the participant a poor protocol candidate, in the opinion of the principal investigator
* Post surgical removal of both ovaries
* Postmenopausal women with amenorrhea greater than 12 months
* Previous history of endometrial biopsy, hysteroscopy, dilatation and curettage, or IUD in place within the past 3 months
* Known participation in a concurrent protocol with a pharmacological intervention
* Recent or concurrent use of systemic steroids (i.e. prednisone) within the past four months of initiating study
* Positive serum pregnancy test at baseline evaluation
* Fasting triglycerides level >= 400 mg/dl
* Cholesterol level >= 240 mg/dl
* LDL level >= 160 mg/dl
* HDL level =< 35 mg/dl
* Hypertension that is currently not under good control, in the judgement of the principal investigator

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2002-02; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change in potential SEBs relevant to endometrial carcinogenesis. | From baseline to completion of hormone therapy

SECONDARY OUTCOMES:
Changes in histology and ultrasound appearance of the endometrium in women with HNPCC | From baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Lu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States